CLINICAL TRIAL: NCT02620241
Title: Influence of Intrapulmonary Percussive Ventilation (IPV) on Gastro-oesophageal Reflux (GOR) in Infants
Brief Title: Influence of Intrapulmonary Percussive Ventilation (IPV) on Gastro-oesophageal Reflux (GOR).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Filip Van Ginderdeuren, FVanGinderdeuren, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VrijeUB
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Gastro-oesophageal Reflux
Keywords: gastro-oesophageal reflux; intrapulmonary percussive ventilation; positioning
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Sitting Position

ARMS (1):
- sitting position (Other): infants are in a sitting position for 20 minutes
  Interventions: Other: sitting position

INTERVENTIONS:
Other: sitting position

SUMMARY:
The study evaluates the effect on gastro-oesophageal reflux (GOR) of infants sitting in a stable upright position during 20 min. This is an addendum to the previous study with record number clinical trials.gov NCT02124863

ELIGIBILITY:
Inclusion Criteria:

* Each child under the age of one year that was referred for 24h pH-MII monitoring to exclude pathological gastro-oesophageal reflux (GOR)

Exclusion Criteria:

* : prematurity (gestational age less than 37 weeks), the use of anti-reflux medication and reflux surgery (Nissen fundoplication)

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
number of reflux episodes | 20 minutes
  number of reflux episodes is counted over 20 min period of time

CONTACTS AND LOCATIONS:
Locations (1):
- UZBrussel, Jette, Brussels Capital, Belgium